CLINICAL TRIAL: NCT03641547
Title: A Phase 1 Dose Escalation Safety Study Combining the ATR Inhibitor M6620 With Chemoradiotherapy in Oesophageal Cancer & Other Solid Cancers Using Time to Event Continual Reassessment Method
Brief Title: M6620 Plus Standard Treatment in Oesophageal and Other Cancer
Acronym: CHARIOT
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Oxford (Other)
Collaborators: Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OCTO_072
Record Dates: First submitted 2018-07-10; First posted 2018-08-22 (Actual); Results first posted 2024-07-18 (Actual); Last update posted 2024-07-18 (Actual); Status verified 2022-04

CONDITIONS: Oesophageal Adenocarcinoma; Squamous Cell Carcinoma; Solid Tumor
Keywords: Oesophageal cancer
MeSH Terms: conditions — Adenocarcinoma Of Esophagus; Carcinoma, Squamous Cell; Esophageal Neoplasms | interventions — Cisplatin; Capecitabine; Radiotherapy

STUDY DESIGN:
Intervention Model Description: CHARIOT will use a single arm, open-label, dose escalation, Time-To-Event Continual Reassessment Method (TiTE-CRM) to find the optimal treatment schedule.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Stage A1, A2 & B (Experimental): The trial is a single arm study. Different populations are recruited to each stage and the stages run independently of each other. Stage A1 & A2 will commence before Stage B so that safety data can be obtained in the palliative setting prior to Stage B commencing. Stage A1 may be ongoing when Stage B begins. Each Stage has a separate eligibility criteria.
  Stage A1: M6620 & palliative radiotherapy Stage A2: M6620 & palliative chemotherapy (Cisplatin & Capecitabine) Stage B: M6620 & definitive chemoradiotherapy
  Interventions: Drug: M6620; Drug: Cisplatin; Drug: Capecitabine; Radiation: Radiotherapy

INTERVENTIONS:
Drug: M6620 — M6620 is an unlicensed small molecule ATR inhibitor which can be used in combination with DNA damaging agents. In pre-clinical models it has substantial activity when given with DNA damaging drugs or ionising radiation. The clinical agent (M6620) is currently studied in a phase I trial in Oxford and other centres in combination with gemcitabine, cisplatin, gemcitabine/cisplatin and cisplatin/etoposide.
Drug: Cisplatin — Cisplatin is a platinum based chemotherapy drug licensed to treat a number of different types of cancer. Cisplatin use is not considered standard practice in Stage A2 & B, therefore Cisplatin is considered an investigational medicinal product for the purpose of this trial.
Drug: Capecitabine — Capecitabine is a chemotherapy drug licensed to treat a number of different types of cancer, it is a noncytotoxic pre-cursor of the cytotoxic 5-fluourouracil. Capecitabine use is not considered standard practice in Stage A2 & B, therefore Capecitabine is considered an investigational medicinal product for the purpose of this trial.
Radiation: Radiotherapy — Stage A1 uses palliative radiotherapy. Stage B uses definitive radiotherapy.

SUMMARY:
This Phase I study will test the combination of a novel ATR inhibitor (M6620) with chemoradiotherapy in oesophageal cancer; utilizing three experimental cohorts (Stage A1, A2 and B).

DETAILED DESCRIPTION:
There is strong scientific rationale for combining ATR inhibitors with DNA damaging agents such as radiation and cisplatin. In particular, ATR inhibition has been shown to be cytotoxic to tumor cells with an impaired DNA damage response, such as those with deficiency in the ATM- or p53 pathway. The high incidence of p53 mutations and the fact that cisplatin and radiation are key therapeutics, makes oesophageal cancer an attractive tumor type to test the activity of an ATR inhibitor. Given the reported synthetic lethal relationship between ATM and ATR, it is likely that ATR inhibition in an ATM- or p53- deficient background will offer a specific and effective way of targeting OAC and SCC of the oesophagus, and enhance the current standard of care.

The trial will be divided into three stages. Stage A1 will explore the combination of M6620 plus radiotherapy in the palliative setting and Stage A2 will explore the combination of M6620 plus chemotherapy in the palliative setting. Stage B, will explore the combination of all 3 (M6620 plus chemoradiotherapy in the radical setting).

In Stage A1 of the study M6620 will be combined with radiotherapy for the first time and the starting dose will be 140mg/m2 M6620, which has been well-tolerated. M6620 will be administered with daily palliative radiotherapy during this stage in order to study the specific interaction of M6620 with radiotherapy (acting as the DNA damaging agent during this trial stage).

In Stage A2 of the study, M6620 will be combined with Cisplatin and Capecitabine combination chemotherapy for the first time; with a starting dose of 90mg/m2 M6620. M6620 will be administered 24 hours post cisplatin infusion, aiming to achieve maximum treatment benefit. Stage A1 and A2 together will help give an indication of a toxicity profile before administration with chemoradiotherapy (Stage B).

ELIGIBILITY:
INCLUSION CRITERIA:

For Stage A1:

1. Histologically confirmed adenocarcinoma or squamous cell carcinoma of the oesophagus (not including cervical oesophagus)
2. Tumor length 15cm or less
3. Any stage of disease that is unsuitable for radical CRT or surgery but suitable for palliative RT
4. Baseline investigations available: staging CT scan (within 42 days before first study dose) and endoscopy
5. Previous chemotherapy treatment completed 28 days before first study dose
6. No oesophageal stent in-situ
7. Any gender, aged ≥16 years.
8. Life expectancy of at least 12 weeks
9. ECOG performance score of 0-1
10. Able to comply with protocol fully - absence of any physical, psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule; those conditions should be discussed with the patient before registration in the trial
11. Able to give written (signed and dated) informed consent according to GCP before registration
12. Hematological and biochemical indices within the ranges below:

    * Haemoglobin: ≥8.0g/dL
    * Platelet count : ≥100x10^9/L
    * Absolute neutrophil count: ≥1.5x10^9/L
    * Total bilirubin: ≤1.5 x upper limit of normal unless the subject has known or suspected Gilbert's syndrome
    * AST/ALT: ≤2.5 times the upper limit of normal; ≤5 times if liver metastases
    * Estimated glomerular filtration rate: ≥40ml/min

For Stage A2:

1. Any histologically confirmed advanced solid tumor that is metastatic or unresectable where Investigator considers Cisplatin and Capecitabine based regimen as appropriate.
2. Baseline investigations available: staging CT scan (within 35 days before first study dose)
3. Previous chemotherapy treatment completed 28 days before first study dose
4. Any gender, aged ≥16 years
5. Life expectancy of at least 12 weeks
6. ECOG performance score of 0-1
7. Able to comply with protocol fully - absence of any physical, psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule; those conditions should be discussed with the patient before registration in the trial
8. Able to give written (signed and dated) informed consent according to GCP before registration
9. Hematological and biochemical indices within the ranges below:

   * Haemoglobin: ≥10.0g/dL
   * Platelet count : ≥100x10^9/L
   * Absolute neutrophil count: ≥1.5x10^9/L
   * Total bilirubin: ≤1.5 x upper limit of normal unless the subject has known or suspected Gilbert's syndrome
   * AST/ALT: ≤2.5 times the upper limit of normal; ≤5 times if liver metastases
   * Ca, Mg, Phosphate: within normal limits
   * Estimated glomerular filtration rate: ≥60ml/min

For Stage B:

1. Histologically confirmed adenocarcinoma or squamous cell carcinoma of the oesophagus including Siewert type 1 or 2 tumors with ≤2cm gastric mucosal extension (not including cervical oesophagus)
2. Tumor length 7cm or less
3. Suitable for radical CRT and surgery not an option due to being medically unfit or unsuitable for surgery or patient choice
4. No oesophageal stent in-situ
5. Endoscopically or radiologically documented measurable disease
6. Diagnostic PET CT scan*
7. Staging CT scan*

   *either CT or PET CT scan within 42 days of first study dose
8. Adequate respiratory and cardiac function tests for safe delivery of CRT in the opinion of the Principle Investigator, specifically cardiac ejection fraction ≥60% and lung function FEV1>1 litre or 40% of predicted value or KCO (DLCO/VA) >40% predicted value.
9. Any gender, aged ≥16 years
10. ECOG performance score of 0-1
11. Able to comply with protocol fully - absence of any physical, psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule; those conditions should be discussed with the patient before registration in the trial
12. Able to give written (signed and dated) informed consent according to GCP before registration
13. Haematological and biochemical indices within the ranges below:

    * Haemoglobin: ≥10.0g/dL
    * Platelet count : ≥100x10^9/L
    * Absolute neutrophil count: ≥1.5x10^9/L
    * Total bilirubin: ≤1.5 x upper limit of normal unless the subject has known or suspected Gilbert's syndrome
    * AST/ALT: ≤2.5 times the upper limit of normal; ≤5 times if liver metastases
    * Ca, Mg, Phosphate: within normal limits
    * Estimated glomerular filtration rate: ≥60ml/min

EXCLUSION CRITERIA:

1. Pregnant or breast-feeding women, or women of childbearing potential unless highly effective contraception is used
2. Untreated and multiple brain metastases
3. Clinically significant cardiovascular event within 6 months before study entry to include: a) congestive heart failure requiring therapy, b) unstable angina pectoris, c) myocardial infarction, d) class II/III/IV cardiac disease (New York Heart Association), e) presence of severe valvular heart disease, f) presence of ventricular arrhythmia requiring treatment
4. History of arrhythmia that is symptomatic or requires treatment (CTCAE 3), symptomatic or uncontrolled atrial fibrillation, despite treatment, or asymptomatic sustained ventricular tachycardia. Subjects with atrial fibrillation controlled by medication are permitted.
5. Uncontrolled hypertension (blood pressure ≥160/100 despite optimal therapy)
6. Second or third degree heart block with or without symptoms
7. QTc >450msec in adult male and >470 msec in adult females (by Fridericia's correction) not due to electrolyte abnormality and that does not resolve with correction of electrolytes.
8. History of congenital long QT syndrome
9. History of torsades de pointes (or any concurrent medication with a known risk of inducing torsades de pointes)
10. Trachea-oesophageal fistula or invasion of the tracheo-bronchial tree
11. Treatment with any other investigational agent, or participation in another clinical trial within 28 days prior to the start of treatment
12. Strong CYP3A inhibitors and inducers or haemopoietic growth factors within 14 days before first dose of M6620 (Berzosertib)
13. HER2 gastro-oesophageal positive cancer where anti-Her2 therapies may be more appropriate (however patients who have failed anti-HER2 therapy may be eligible for stage A1 and A2)
14. Unable to have or unwilling to change to low molecular weight heparin instead of Warfarin
15. Other psychological, social or medical condition, physical examination finding or a laboratory abnormality that the Investigator considers would make the patient a poor trial candidate or could interfere with protocol compliance or the interpretation of trial results.
16. Any other active malignancy, with the exception of adequately treated cone-biopsied in situ carcinoma of the cervix uteri and non-melanoma skin lesions.
17. Patients who are known to be serologically positive for Hepatitis B, Hepatitis C or HIV.

Additional Exclusion Criteria for Stage A1 and B:

1) Previous radiotherapy to thorax or upper abdomen

Additional exclusion criteria for Stage A2 and B:

1. History of hand-foot syndrome
2. History of hearing impairment
3. Live vaccine received within 30 days prior to treatment start
4. Complete or Partial DPD deficiency

Additional Exclusion Criteria for Stage B:

1) Previous chemotherapy

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2018-12-04 (Actual); Primary Completion 2022-04-04 (Actual); Study Completion 2022-04-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Maria A Hawkins, MD FRCR MRCP, Principal Investigator — University College, London
Locations (5):
- United Kingdom (5):
  - Velindre Cancer Centre, Cardiff
  - Beatson Cancer Centre, Glasgow
  - St James's University Hospital, Leeds
  - The Christie, Manchester
  - The Churchill Hospital, Oxford University Hospitals Trust, Oxford

REFERENCES:
- [Derived] Javed SR, Lord S, El Badri S, Harman R, Holmes J, Kamzi F, Maughan T, McIntosh D, Mukherjee S, Ooms A, Radhakrishna G, Shaw P, Hawkins MA. CHARIOT: a phase I study of berzosertib with chemoradiotherapy in oesophageal and other solid cancers using time to event continual reassessment method. Br J Cancer. 2024 Feb;130(3):467-475. doi: 10.1038/s41416-023-02542-1. Epub 2023 Dec 21. PMID 38129525
- [Derived] van Werkhoven E, Hinsley S, Frangou E, Holmes J, de Haan R, Hawkins M, Brown S, Love SB. Practicalities in running early-phase trials using the time-to-event continual reassessment method (TiTE-CRM) for interventions with long toxicity periods using two radiotherapy oncology trials as examples. BMC Med Res Methodol. 2020 Jun 22;20(1):162. doi: 10.1186/s12874-020-01012-z. PMID 32571298

RESULTS

PARTICIPANT FLOW:
Groups:
- A1 - Dose Level 1: Radiotherapy + M6620 (Berzosertib) administered at 140 mg/m2 on days 2, 9, 16.
- A1 - Dose Level 2: Radiotherapy + M6620 (Berzosertib) administered at 140 mg/m2 on days 2, 5, 9, 12, 16.
- A1 - Dose Level 3: Radiotherapy + M6620 (Berzosertib) administered at 140 mg/m2 on days 2, 5, 9, 12, 16, 19.
- A1 - Dose Level 4: Radiotherapy + M6620 (Berzosertib) administered at 240 mg/m2 on days 2, 9, 16.
- A1 - Dose Level 5: Radiotherapy + M6620 (Berzosertib) administered at 240 mg/m2 on days 2, 5, 9, 12, 16.
- A1 - Dose Level 6: Radiotherapy + M6620 (Berzosertib) administered at 240 mg/m2 on days 2, 5, 9, 12, 16, 19.
- A2 - Dose Level 1: Cisplatin/capecitabine + M6620 (Berzosertib) administered at 90 mg/m2 once a week for 18 weeks.
- A2 - Dose Level 2: Cisplatin/capecitabine + M6620 (Berzosertib) administered at 90 mg/m2 twice a week for 18 weeks.
- A2 - Dose Level 3: Cisplatin/capecitabine + M6620 (Berzosertib) administered at 140 mg/m2 once a week for 18 weeks.
- A2 - Dose Level 4: Cisplatin/capecitabine + M6620 (Berzosertib) administered at 140 mg/m2 twice a week for 18 weeks.
Period: Overall Study
Arm/Group | A1 - Dose Level 1 | A1 - Dose Level 2 | A1 - Dose Level 3 | A1 - Dose Level 4 | A1 - Dose Level 5 | A1 - Dose Level 6 | A2 - Dose Level 1 | A2 - Dose Level 2 | A2 - Dose Level 3 | A2 - Dose Level 4
Started | 3 | 1 | 1 | 1 | 1 | 9 | 5 | 1 | 9 | 5
Completed | 3 | 1 | 1 | 1 | 1 | 9 | 2 | 1 | 4 | 3
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 5 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | A1 - Dose Level 1 | A1 - Dose Level 2 | A1 - Dose Level 3 | A1 - Dose Level 4 | A1 - Dose Level 5 | A1 - Dose Level 6 | A2 - Dose Level 1 | A2 - Dose Level 2 | A2 - Dose Level 3 | A2 - Dose Level 4 | Total
Number analyzed (Participants) | 3 | 1 | 1 | 1 | 1 | 9 | 5 | 1 | 9 | 5 | 36
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 2 | 0 | 1 | 0 | 0 | 5 | 2 | 1 | 3 | 3 | 17
  >=65 years | 1 | 1 | 0 | 1 | 1 | 4 | 3 | 0 | 6 | 2 | 19
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 1 | 0 | 1 | 2 | 0 | 6 | 3 | 13
  Male | 3 | 1 | 1 | 0 | 1 | 8 | 3 | 1 | 3 | 2 | 23
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 3 | 1 | 1 | 1 | 1 | 9 | 5 | 1 | 9 | 5 | 36
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Smoking status [Count of Participants; unit: Participants]
  Ex-smoker | 2 | 1 | 1 | 0 | 1 | 6 | 1 | 1 | 4 | 3 | 20
  Never smoked | 1 | 0 | 0 | 1 | 0 | 3 | 3 | 0 | 5 | 2 | 15
  Current smoker | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Locoregional Disease [Count of Participants; unit: Participants]
  Yes | 3 | 1 | 1 | 1 | 1 | 6 | 1 | 0 | 6 | 3 | 23
  No | 0 | 0 | 0 | 0 | 0 | 3 | 4 | 1 | 3 | 2 | 13
Distant Metastases [Count of Participants; unit: Participants]
  Yes | 1 | 0 | 0 | 1 | 0 | 4 | 5 | 1 | 8 | 5 | 25
  No | 2 | 1 | 1 | 0 | 1 | 5 | 0 | 0 | 1 | 0 | 11
Prior Radiotherapy [Count of Participants; unit: Participants]
  Yes | 0 | 0 | 0 | 0 | 0 | 1 | 4 | 0 | 2 | 2 | 9
  No | 3 | 1 | 1 | 1 | 1 | 8 | 1 | 1 | 7 | 3 | 27
Prior Systemic Treatment [Count of Participants; unit: Participants]
  Yes | 2 | 0 | 1 | 1 | 1 | 8 | 4 | 1 | 9 | 5 | 32
  No | 1 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 4
Tumour grade [Count of Participants; unit: Participants]
  Well differentiated (G1) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2
  Moderately differentiated (G2) | 1 | 0 | 0 | 0 | 0 | 2 | 1 | 1 | 3 | 0 | 8
  Poorly differentiated (G3) | 0 | 1 | 1 | 1 | 1 | 4 | 4 | 0 | 0 | 3 | 15
  Unknown or cannot be assessed (GX) | 1 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 5 | 2 | 11

OUTCOME MEASURES:

1. Primary Outcome: STAGE A1 - Number of Dose Limiting Toxicities for M6620 (Berzosertib) Administered Concomitantly With Radiotherapy (RT) in the Palliative Treatment of Oesophageal Cancer.
Description: To determine the best tolerated M6620 (Berzosertib) treatment schedule (or phase II recommended dose, RPTD) administered concomitantly with radiotherapy (RT) only in the palliative treatment of oesophageal cancer.
Time Frame: From start of M6620 (Berzosertib) treatment to 6-week follow up visit (9 weeks)
Measure: Number; unit: Dose Limiting Toxicities (DLTs)
Arm/Group | A1 - Dose Level 1 | A1 - Dose Level 2 | A1 - Dose Level 3 | A1 - Dose Level 4 | A1 - Dose Level 5 | A1 - Dose Level 6
Number analyzed (Participants) | 3 | 1 | 1 | 1 | 1 | 9
Dose Limiting Toxicities (DLTs) | 0 | 0 | 0 | 0 | 0 | 0
Statistical Analysis 1: Comparison: A1 - Dose Level 1 vs A1 - Dose Level 2 vs A1 - Dose Level 3 vs A1 - Dose Level 4 vs A1 - Dose Level 5 vs A1 - Dose Level 6; The primary analysis is performed using the Time-To-Event Continual Reassessment Method (TiTE-CRM). Giving posterior estimates for the probability of toxicity (DLT) at each dose level; Test type: Other; Post prob of tox at dose level 6 = 0.029, 95% CI 2-sided [0 to 0.165]

2. Primary Outcome: STAGE A2 - Number of Dose Limiting Toxicities for M6620 (Berzosertib) Administered Concomitantly With Chemotherapy (Cisplatin and Capecitabine) in the Palliative Treatment of Solid Cancer.
Description: To determine the best tolerated M6620 (Berzosertib) treatment schedule (or phase II recommended dose, RPTD) administered concomitantly with chemotherapy (cisplatin and capecitabine) only in the palliative treatment of solid cancer.
Time Frame: From start of M6620 (Berzosertib) treatment to end of first week of cycle two of chemotherapy (4 weeks)
Measure: Number; unit: Dose Limiting Toxicities (DLTs)
Arm/Group | A2 - Dose Level 1 | A2 - Dose Level 2 | A2 - Dose Level 3 | A2 - Dose Level 4
Number analyzed (Participants) | 4 | 1 | 9 | 4
Dose Limiting Toxicities (DLTs) | 0 | 0 | 2 | 0
Statistical Analysis 1: Comparison: A2 - Dose Level 1 vs A2 - Dose Level 2 vs A2 - Dose Level 3 vs A2 - Dose Level 4; The primary analysis is performed using the Time-To-Event Continual Reassessment Method (TiTE CRM). Giving posterior estimates for the probability of toxicity (DLT) at each dose level; Test type: Other; Post prob of tox at dose level 4 = 0.185, 95% CI 2-sided [0.042 to 0.397]

3. Primary Outcome: STAGE B - To Determine the Best Tolerated M6620 (Berzosertib) Treatment Schedule (or RPTD) Administered Concomitantly With Radiotherapy (dCRT) in Combination With Cisplatin and Capecitabine in the Radical Treatment of Oesophageal Cancer.
Description: Highest treatment schedule resulting in less than 45% dose limiting toxicity (DLT) rate.
Time Frame: 24 weeks
Population: Due to lack of funding, Stage B was not completed.
Groups:
- Stage A1, A2 & B: The trial is a single arm study. Different populations were recruited to each stage and the stages ran independently of each other. Stage A1 & A2 were planned to commence before Stage B so that safety data could be obtained in the palliative setting prior to Stage B commencing. However, due to lack of funding, Stage B was not completed.
  Stage A1: M6620 & palliative radiotherapy Stage A2: M6620 & palliative chemotherapy (Cisplatin & Capecitabine) Stage B: M6620 & definitive chemoradiotherapy
  M6620: M6620 is an unlicensed small molecule ATR inhibitor which can be used in combination with DNA damaging agents. In pre-clinical models it has substantial activity when given with DNA damaging drugs or ionising radiation. The clinical agent (M6620) is currently studied in a phase I trial in Oxford and other centres in combination with gemcitabine, cisplatin, gemcitabine/cisplatin and cisplatin/etoposide.
Arm/Group | Stage A1, A2 & B
Number analyzed (Participants) | 0

4. Secondary Outcome: STAGE A1 - Severity of Worst Adverse Events for M6620 (Berzosertib) Administered Concomitantly With Radiotherapy (RT) in the Palliative Treatment of Oesophageal Cancer.
Description: Toxicity profile when M6620 is administered concomitantly with RT in the palliative treatment of oesophageal cancer. Worst grade adverse event for each patient by dose schedule (according to the Common Terminology Criteria for Adverse Events, Version 4.03). Grade 1 (mild); Grade 2 (moderate); Grade 3 (severe or medically significant, but not immediately life-threatening); Grade 4 (life-threatening); Grade 5 (death).
Time Frame: From start of M6620 (Berzosertib) treatment to 9-week follow up visit (12 weeks)
Measure: Count of Participants; unit: Participants
Arm/Group | A1 - Dose Level 1 | A1 - Dose Level 2 | A1 - Dose Level 3 | A1 - Dose Level 4 | A1 - Dose Level 5 | A1 - Dose Level 6
Number analyzed (Participants) | 3 | 1 | 1 | 1 | 1 | 9
Participants
  Worst AE: Grade 1 | 1 | 1 | 0 | 1 | 1 | 2
  Worst AE: Grade 2 | 2 | 0 | 0 | 0 | 0 | 1
  Worst AE: Grade 3 | 0 | 0 | 1 | 0 | 0 | 6
  Worst AE: Grade 4 | 0 | 0 | 0 | 0 | 0 | 0

5. Secondary Outcome: STAGE A1 - Number of Patients Completing at Least 75%, 90% and 100% of the Planned Treatment Dose of M6620 (Berzosertib) in Combination With Palliative Radiotherapy
Description: Treatment compliance of M6620 (Berzosertib) and palliative radiotherapy when taken concomitantly.
Time Frame: From start of M6620 (Berzosertib) treatment to last dose (3 weeks)
Measure: Count of Participants; unit: Participants
Arm/Group | A1 - Dose Level 1 | A1 - Dose Level 2 | A1 - Dose Level 3 | A1 - Dose Level 4 | A1 - Dose Level 5 | A1 - Dose Level 6
Number analyzed (Participants) | 3 | 1 | 1 | 1 | 1 | 9
Participants
  Radiotherapy compliance: 100% | 3 | 1 | 1 | 1 | 1 | 7
  Radiotherapy compliance: >=90%, <100% | 0 | 0 | 0 | 0 | 0 | 2
  Radiotherapy compliance: >=75%,<90% | 0 | 0 | 0 | 0 | 0 | 0
  Radiotherapy compliance: <75% | 0 | 0 | 0 | 0 | 0 | 0
  M6620 (Berzosertib) compliance: 100% | 2 | 1 | 0 | 1 | 0 | 5
  M6620 (Berzosertib) compliance: >=90%, <100% | 0 | 0 | 0 | 0 | 0 | 0
  M6620 (Berzosertib) compliance: >=75%,<90% | 1 | 0 | 1 | 0 | 1 | 3
  M6620 (Berzosertib) compliance: <75% | 0 | 0 | 0 | 0 | 0 | 1

6. Secondary Outcome: STAGE A1 - Objective Tumour Response to M6620 (Berzosertib) Plus Radiotherapy, as Evaluated by CT Scan and Quantified by RECIST 1.1.
Description: Efficacy of the combination (M6620 and radiotherapy), measured by objective tumour response via RECIST 1.1 (Eisenhauer EA, Therasse P, Bogaerts J, et al. New response evaluation criteria in solid tumours: revised RECIST guideline (version 1.1). Eur J Cancer. 2009;45(2):228-247. doi:10.1016/j.ejca.2008.10.026). From Progressive Disease (PD) to Complete Response (CR).
Time Frame: At 12 weeks following start of M6620 (Berzosertib) treatment
Population: Overall RECIST at 12 Weeks
Measure: Count of Participants; unit: Participants
Arm/Group | A1 - Dose Level 1 | A1 - Dose Level 2 | A1 - Dose Level 3 | A1 - Dose Level 4 | A1 - Dose Level 5 | A1 - Dose Level 6
Number analyzed (Participants) | 3 | 1 | 1 | 1 | 1 | 9
Participants
  Complete Response | 0 | 0 | 0 | 0 | 0 | 0
  Partial Response | 1 | 0 | 0 | 0 | 0 | 1
  Stable Disease | 1 | 1 | 1 | 1 | 0 | 2
  Progressive Disease | 0 | 0 | 0 | 0 | 1 | 2
  Not Evaluable | 0 | 0 | 0 | 0 | 0 | 1
  Missing Data | 1 | 0 | 0 | 0 | 0 | 3

7. Secondary Outcome: STAGE A2 - Severity of Worst Adverse Events for M6620 (Berzosertib) Administered Concomitantly With Chemotherapy (Cisplatin and Capecitabine) in the Palliative Treatment of Solid Cancer
Description: Toxicity profile when M6620 is administered concomitantly with chemotherapy in the treatment of oesophageal cancer. Worst grade adverse event for each patient by dose schedule (according to the Common Terminology Criteria for Adverse Events, Version 4.03). Grade 1 (mild); Grade 2 (moderate); Grade 3 (severe or medically significant, but not immediately life-threatening); Grade 4 (life-threatening); Grade 5 (death).
Time Frame: From start of M6620 (Berzosertib) treatment to 8-week post-end of treatment follow up visit (26 weeks)
Population: 2 participants were not included in this analysis as they did not take any IMP.
Measure: Count of Participants; unit: Participants
Arm/Group | A2 - Dose Level 1 | A2 - Dose Level 2 | A2 - Dose Level 3 | A2 - Dose Level 4
Number analyzed (Participants) | 4 | 1 | 9 | 4
Participants
  Worst AE: Grade 1 | 0 | 0 | 0 | 0
  Worst AE: Grade 2 | 2 | 1 | 2 | 1
  Worst AE: Grade 3 | 1 | 0 | 6 | 2
  Worst AE: Grade 4 | 1 | 0 | 1 | 1

8. Secondary Outcome: STAGE A2 - Number of Patients Completing at Least 75%, 90% and 100% of the Planned Treatment Dose of M6620 (Berzosertib) in Combination With Chemotherapy (Cisplatin and Capecitabine) in the Palliative Treatment of Solid Cancer.
Description: Treatment compliance of M6620 (Berzosertib), capecitabine and cisplatin when taken concomitantly.
Time Frame: From start of M6620 (Berzosertib) treatment to last dose (18 weeks)
Population: 2 participants were not included in this analysis as they did not take any IMP.
Measure: Count of Participants; unit: Participants
Arm/Group | A2 - Dose Level 1 | A2 - Dose Level 2 | A2 - Dose Level 3 | A2 - Dose Level 4
Number analyzed (Participants) | 4 | 1 | 9 | 4
Participants
  Capecitabine compliance: 100% | 0 | 0 | 1 | 0
  Capecitabine compliance: >=90%, <100% | 1 | 0 | 0 | 0
  Capecitabine compliance: >=75%, <90% | 0 | 1 | 0 | 0
  Capecitabine compliance: <75% | 3 | 0 | 8 | 4
  Cisplatin compliance: 100% | 1 | 0 | 2 | 0
  Cisplatin compliance: >=90%, <100% | 0 | 0 | 1 | 0
  Cisplatin compliance: >=75%, <90% | 0 | 1 | 0 | 0
  Cisplatin compliance: <75% | 3 | 0 | 6 | 4
  M6620 (Berzosertib) compliance in cycle 1: 100% | 3 | 0 | 4 | 2
  M6620 (Berzosertib) compliance in cycle 1: >=90%, <100% | 0 | 0 | 0 | 0
  M6620 (Berzosertib) compliance in cycle 1: >=75%, <90% | 0 | 1 | 0 | 0
  M6620 (Berzosertib) compliance in cycle 1: <75% | 1 | 0 | 5 | 2

9. Secondary Outcome: STAGE A2 - Objective Tumour Response to M6620 (Berzosertib) Plus Chemotherapy, as Evaluated by CT Scan and Quantified by RECIST 1.1.
Description: Efficacy of the combination (M6620 and chemotherapy), measured by objective tumour response via RECIST 1.1 (Eisenhauer EA, Therasse P, Bogaerts J, et al. New response evaluation criteria in solid tumours: revised RECIST guideline (version 1.1). Eur J Cancer. 2009;45(2):228-247. doi:10.1016/j.ejca.2008.10.026). From Progressive Disease (PD) to Complete Response (CR).
Time Frame: At 12 weeks following start of M6620 (Berzosertib) treatment
Population: Overall RECIST at 12 Weeks
Measure: Count of Participants; unit: Participants
Arm/Group | A2 - Dose Level 1 | A2 - Dose Level 2 | A2 - Dose Level 3 | A2 - Dose Level 4
Number analyzed (Participants) | 5 | 1 | 9 | 5
Participants
  Complete Response | 0 | 0 | 0 | 0
  Partial Response | 1 | 1 | 0 | 1
  Stable Disease | 0 | 0 | 2 | 2
  Progressive Disease | 0 | 0 | 1 | 0
  Not Evaluable | 0 | 0 | 0 | 0
  Missing Data | 4 | 0 | 6 | 2

10. Secondary Outcome: STAGE B - To Determine the Safety and Toxicity Profile of M6620 (Berzosertib) Administered Concomitantly With dCRT in Combination With Cisplatin and Capecitabine in the Radical Treatment of Oesophageal Cancer.
Description: Any toxicity grade ≥3 graded according to CTCAE v4.03 and length of time for toxicity to resolve.
Time Frame: 24 weeks
Population: Due to lack of funding, Stage B was not completed.
Groups:
- Stage A1, A2 & B: The trial was a single arm study. Different populations were recruited to each stage and the stages ran independently of each other. Stage A1 & A2 were planned to commence before Stage B so that safety data could be obtained in the palliative setting prior to Stage B commencing. However, Stage B did not go ahead due to lack of funding. Each Stage has a separate eligibility criteria.
  Stage A1: M6620 & palliative radiotherapy Stage A2: M6620 & palliative chemotherapy (Cisplatin & Capecitabine) Stage B: M6620 & definitive chemoradiotherapy
  M6620: M6620 is an unlicensed small molecule ATR inhibitor which can be used in combination with DNA damaging agents. In pre-clinical models it has substantial activity when given with DNA damaging drugs or ionising radiation. The clinical agent (M6620) is currently studied in a phase I trial in Oxford and other centres in combination with gemcitabine, cisplatin, gemcitabine/cisplatin and cisplatin/etoposide.
Arm/Group | Stage A1, A2 & B
Number analyzed (Participants) | 0

11. Secondary Outcome: STAGE B - To Determine Tolerance and Ability to Deliver M6620 (Berzosertib) in Combination With Standard dCRT.
Description: Treatment tolerance and deliverability measured by proportion of patients completing at least 80% of the planned chemotherapy dose and at least 20 fractions of RT.
Time Frame: 24 weeks
Population: Due to lack of funding, Stage B was not completed.
Arm/Group | Stage A1, A2 & B
Number analyzed (Participants) | 0

12. Secondary Outcome: STAGE B - To Determine the Efficacy of the Long Term Safety of the Treatment Combination.
Description: To measure objective tumour response as evaluated by CT scan and quantified by RECIST 1.1 and endoscopic biopsy findings & PFS and OS from D1
Time Frame: 24 weeks
Population: Due to lack of funding, Stage B was not completed.
Arm/Group | Stage A1, A2 & B
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Stage A1 - adverse events (including serious) are reported from start of M6620 (Berzosertib) treatment to follow up visit at 9 weeks post-end of treatment (12 weeks). Stage A2 - adverse events (including serious) are reported from start of M6620 (Berzosertib) treatment to follow up visit at 8 weeks post-end of treatment (26 weeks). Both Stages - Mortality is reported from start of M6620 (Berzosertib) treatment to patient completion of trial at 12 months after start of treatment (12 months).
Arm/Group | A1 - Dose Level 1 | A1 - Dose Level 2 | A1 - Dose Level 3 | A1 - Dose Level 4 | A1 - Dose Level 5 | A1 - Dose Level 6 | A2 - Dose Level 1 | A2 - Dose Level 2 | A2 - Dose Level 3 | A2 - Dose Level 4
All-Cause Mortality (participants affected / at risk) | 1/3 | 1/1 | 0/1 | 1/1 | 1/1 | 5/9 | 3/5 | 1/1 | 5/9 | 2/5
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/1 | 0/1 | 0/1 | 0/1 | 2/9 | 0/5 | 0/1 | 3/9 | 0/5
Other Adverse Events (participants affected / at risk) | 3/3 | 1/1 | 1/1 | 1/1 | 1/1 | 9/9 | 4/5 | 1/1 | 9/9 | 4/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | A1 - Dose Level 1 (N=3) | A1 - Dose Level 2 (N=1) | A1 - Dose Level 3 (N=1) | A1 - Dose Level 4 (N=1) | A1 - Dose Level 5 (N=1) | A1 - Dose Level 6 (N=9) | A2 - Dose Level 1 (N=5) | A2 - Dose Level 2 (N=1) | A2 - Dose Level 3 (N=9) | A2 - Dose Level 4 (N=5)
Gastrostomy tube site complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Rig accidentally fallen out
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | A1 - Dose Level 1 (N=3) | A1 - Dose Level 2 (N=1) | A1 - Dose Level 3 (N=1) | A1 - Dose Level 4 (N=1) | A1 - Dose Level 5 (N=1) | A1 - Dose Level 6 (N=9) | A2 - Dose Level 1 (N=5) | A2 - Dose Level 2 (N=1) | A2 - Dose Level 3 (N=9) | A2 - Dose Level 4 (N=5)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vascular disorders (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 4 (5) | 0 (0)
General disorders and administration site conditions (General disorders) | 2 (4) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 4 (5) | 3 (6) | 1 (1) | 5 (13) | 4 (23)
Reproductive system and breast disorders (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Respiratory, thoracic and mediastinal disorders (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (2) | 1 (1) | 1 (1) | 1 (2) | 3 (4) | 2 (5) | 1 (2) | 2 (2) | 3 (5)
Psychiatric disorders (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Investigations (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (7) | 1 (1) | 1 (2) | 5 (21) | 1 (1)
Injury, poisoning and procedural complications (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Nervous system disorders (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (5) | 1 (2) | 0 (0) | 1 (1) | 3 (3)
Blood and lymphatic system disorders (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (5) | 2 (5) | 1 (2) | 6 (14) | 3 (17)
Ear and labyrinth disorders (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (5)
Eye disorders (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Gastrointestinal disorders (Gastrointestinal disorders) | 2 (3) | 1 (1) | 1 (3) | 0 (0) | 1 (1) | 8 (20) | 2 (4) | 0 (0) | 6 (15) | 4 (20)
Hepatobiliary disorders (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin and subcutaneous tissue disorders (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 5 (13) | 0 (0) | 1 (1) | 1 (8) | 2 (3)
Renal and urinary disorders (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Musculoskeletal and connective tissue disorders (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 2 (2) | 0 (0) | 1 (3) | 3 (4) | 3 (6)
Infections and infestations (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 3 (7) | 1 (6) | 4 (4) | 2 (3)
Metabolism and nutrition disorders (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 5 (6) | 1 (2) | 1 (1) | 5 (8) | 3 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-10-26): https://cdn.clinicaltrials.gov/large-docs/47/NCT03641547/Prot_000.pdf
  • Statistical Analysis Plan (2021-01-07): https://cdn.clinicaltrials.gov/large-docs/47/NCT03641547/SAP_001.pdf